CLINICAL TRIAL: NCT03130868
Title: Microbiome Changes in Severe Burns
Acronym: Microbiome
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A16-761
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Burns Greater Than 20% BSAB; Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fecal samples from patients will be non-invasively collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Characterizing changes in the microbiome — Analyzing the microbial content from stool samples

SUMMARY:
The purpose of the study is characterizing changes in the microbiome of severely-injured adult patients as they progress through stages of injury, reconstruction, and recovery from burns.

DETAILED DESCRIPTION:
There exists a vast collection of bacteria that live on, and within, each human body. All surfaces exposed to the external environment, such as the nares, mouth, airway, skin, and intestines, are colonized, and it is estimated that over 100 trillion microbes live within the gastrointestinal tract alone. The interactions between these colonizers and their host have been demonstrated to affect myriad aspects of human health from autism and inflammatory bowel disease to cancer therapy response. Investigations into the role of the intestinal microbiome in sepsis have been ongoing for decades. Data has shown that critically ill patients can not only experience increased intestinal permeability - a factor that allows for the translocation of bacteria and non-microbial tissue injurious factors into the, primarily lymphatic, circulation, but also a disruption of the symbiotic relationship to one of dysbiosis, resulting in what is known as a "pathobiome."

That the microbiome is affected by thermal injury should be no surprise; burn injury has been shown to drive significant intestinal ischemia and inflammation with subsequently increased intestinal permeability. , Burn-induced lung injury has been linked to these changes, and alterations in the microbiome between critically-burned patients (when compared with healthy controls) have been demonstrated, with resultant overgrowth of gram-negative anaerobes. Thus, the microbiome has a clear role in affecting the clinical course of thermally-injured patients.

This is a descriptive case series study examining microbiome changes in two adult patients admitted with severe burn injuries. This will be done by obtaining regular stool samples and analyzing the microbial content, as well as obtaining clinical data on patients including those factors likely to influence the microbial content.

ELIGIBILITY:
Inclusion Criteria:

* sustained greater than or equal to 20% body surface area of the body (BSAB)

Exclusion Criteria:

* pre-existing clinical infections
* historical evidence of gastrointestinal disease such as Ulcerative Colitis
* Crohn's disease
* Celiac disease
* historical evidence of gastrointestinal Clostridium difficile infection
* no anti-biotic use for 3 months prior to admission
* AIDS
* immune suppressing medications or metastasized cancer
* peritonitis
* non English-speaking

Ages: 17 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will be admitted patients at the Regions Hospital Burn Center
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
microbial diversity of stool samples | up to 6 months
  We will be analyzing the stool composition at the phyla level, looking at the percentages of the five major phyla - Firmicutes, Bacteroidetes, Proteobacteria, Acitonobacteria, and Fusobacteria

CONTACTS AND LOCATIONS:
Overall Officials: William J Mohr, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Round JL, Mazmanian SK. The gut microbiota shapes intestinal immune responses during health and disease. Nat Rev Immunol. 2009 May;9(5):313-23. doi: 10.1038/nri2515. PMID 19343057
- [Background] Clemente JC, Ursell LK, Parfrey LW, Knight R. The impact of the gut microbiota on human health: an integrative view. Cell. 2012 Mar 16;148(6):1258-70. doi: 10.1016/j.cell.2012.01.035. PMID 22424233
- [Background] Vetizou M, Pitt JM, Daillere R, Lepage P, Waldschmitt N, Flament C, Rusakiewicz S, Routy B, Roberti MP, Duong CP, Poirier-Colame V, Roux A, Becharef S, Formenti S, Golden E, Cording S, Eberl G, Schlitzer A, Ginhoux F, Mani S, Yamazaki T, Jacquelot N, Enot DP, Berard M, Nigou J, Opolon P, Eggermont A, Woerther PL, Chachaty E, Chaput N, Robert C, Mateus C, Kroemer G, Raoult D, Boneca IG, Carbonnel F, Chamaillard M, Zitvogel L. Anticancer immunotherapy by CTLA-4 blockade relies on the gut microbiota. Science. 2015 Nov 27;350(6264):1079-84. doi: 10.1126/science.aad1329. Epub 2015 Nov 5. PMID 26541610
- [Background] Carrico CJ, Meakins JL, Marshall JC, Fry D, Maier RV. Multiple-organ-failure syndrome. Arch Surg. 1986 Feb;121(2):196-208. doi: 10.1001/archsurg.1986.01400020082010. No abstract available. PMID 3484944
- [Background] Deitch EA. Gut-origin sepsis: evolution of a concept. Surgeon. 2012 Dec;10(6):350-6. doi: 10.1016/j.surge.2012.03.003. Epub 2012 Apr 23. PMID 22534256
- [Background] Krezalek MA, DeFazio J, Zaborina O, Zaborin A, Alverdy JC. The Shift of an Intestinal "Microbiome" to a "Pathobiome" Governs the Course and Outcome of Sepsis Following Surgical Injury. Shock. 2016 May;45(5):475-82. doi: 10.1097/SHK.0000000000000534. PMID 26863118
- [Background] Honda K, Littman DR. The microbiome in infectious disease and inflammation. Annu Rev Immunol. 2012;30:759-95. doi: 10.1146/annurev-immunol-020711-074937. Epub 2012 Jan 6. PMID 22224764
- [Background] Jakobsson HE, Rodriguez-Pineiro AM, Schutte A, Ermund A, Boysen P, Bemark M, Sommer F, Backhed F, Hansson GC, Johansson ME. The composition of the gut microbiota shapes the colon mucus barrier. EMBO Rep. 2015 Feb;16(2):164-77. doi: 10.15252/embr.201439263. Epub 2014 Dec 18. PMID 25525071